CLINICAL TRIAL: NCT04946825
Title: A Randomized Controlled Trial of Smoking Cessation Treatment for Young Adult Dual Users of Combustible and Electronic Cigarettes
Brief Title: Quit Smoking Study for People Who Use E-Cigarettes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Elias Klemperer, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001059
Record Dates: First submitted 2021-06-10; First posted 2021-07-01 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Nicotine Addiction; E-Cig Use; Quitting Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Quit cigarettes, but continue using e-cigarettes, with nicotine replacement therapy and text support (Experimental): Participants in this arm will be instructed to quit tobacco cigarettes with nicotine replacement therapy (patches and lozenges) and text message support. In addition, these participants will be encouraged to continue using electronic cigarettes to help them quit smoking tobacco cigarettes.
  Interventions: Drug: Nicotine replacement therapy patch; Drug: Nicotine replacement therapy lozenge; Behavioral: Continue electronic cigarettes
- Quit cigarettes and quit e-cigarettes with nicotine replacement therapy and text support. (Experimental): Participants in this arm will be instructed to quit tobacco cigarettes and quit electronic cigarettes with nicotine replacement therapy (patches and lozenges) and text message support.
  Interventions: Drug: Nicotine replacement therapy patch; Drug: Nicotine replacement therapy lozenge; Behavioral: Quit electronic cigarettes
- Quit cigarettes, but continue using e-cigarettes, with text support. (Experimental): Participants in this arm will be instructed to quit tobacco cigarettes with text message support. In addition, these participants will be encouraged to continue using electronic cigarettes to help them quit smoking tobacco cigarettes.
  Interventions: Behavioral: Continue electronic cigarettes
- Quit cigarettes and quit e-cigarettes with text support. (Experimental): Participants in this arm will be instructed to quit tobacco cigarettes and quit electronic cigarettes with text message support.
  Interventions: Behavioral: Quit electronic cigarettes

INTERVENTIONS:
Drug: Nicotine replacement therapy patch — The nicotine patch is attached to the participant's skin and provides a slight constant stream of nicotine. The smaller dose is meant to reduce nicotine dependence.
  Arms: Quit cigarettes and quit e-cigarettes with nicotine replacement therapy and text support.; Quit cigarettes, but continue using e-cigarettes, with nicotine replacement therapy and text support
Drug: Nicotine replacement therapy lozenge — The nicotine lozenge contains small amounts of nicotine, which a participant slowly dissolves in their mouth. Like the patch, the smaller dose is meant to reduce nicotine dependence.
  Arms: Quit cigarettes and quit e-cigarettes with nicotine replacement therapy and text support.; Quit cigarettes, but continue using e-cigarettes, with nicotine replacement therapy and text support
Behavioral: Quit electronic cigarettes — Participants will receive instruction and text message support to quit electronic cigarettes when they quit combustible cigarettes.
  Arms: Quit cigarettes and quit e-cigarettes with nicotine replacement therapy and text support.; Quit cigarettes and quit e-cigarettes with text support.
Behavioral: Continue electronic cigarettes — Participants will receive instruction and text message support to continue using electronic cigarettes after they quit combustible cigarettes.
  Arms: Quit cigarettes, but continue using e-cigarettes, with nicotine replacement therapy and text support; Quit cigarettes, but continue using e-cigarettes, with text support.

SUMMARY:
The overarching aim of this proposed randomized controlled trial (RCT) is to test nicotine replacement therapy (NRT) with text message support for two smoking cessation approaches among young adult dual users of combustible cigarettes (CC) and electronic cigarettes (EC). The investigators will use a 2x2 factorial design to randomize 390 participants to receive A) NRT plus text messages to quit CCs only, B) NRT plus text messages to quit CCs and ECs simultaneously, C) text messages alone to quit CCs only, or D) text messages alone to quit CCs and ECs simultaneously. The investigators primary outcome will be 7-day point-prevalence abstinence at the end of treatment (i.e., 3 months after randomization). The investigators will recruit participants using national advertising strategies. All treatment will be provided remotely in order to increase treatment access and comply with current COVID-19 restrictions.

DETAILED DESCRIPTION:
The overarching aim of this proposed randomized controlled trial (RCT) is to test nicotine replacement therapy (NRT) with text message support for two smoking cessation approaches among young adult dual users of ombustible cigarettes (CC) and electronic cigarettes (EC). The investigators will use a 2x2 factorial design (Table 1) to randomize 390 participants to receive A) NRT plus text messages to quit CCs only, B) NRT plus text messages to quit CCs and ECs simultaneously, C) text messages alone to quit CCs only, or D) text messages alone to quit CCs and ECs simultaneously. The investigators' primary outcome will be 7-day point-prevalence abstinence at the end of treatment (i.e., 3 months after randomization). All treatment will be provided remotely in order to increase treatment access and comply with COVID-19 restrictions. The proposed RCT addresses the following specific aims:

Aim 1: To test whether NRT is an effective smoking cessation treatment for young adult dual users of ECs and CCs.

Aim 2: To identify the influence of continued EC use versus stopping ECs on achieving CC abstinence among young adult dual users of ECs and CCs.

Aim 3: To identify whether continued EC use results in more acute adverse events than stopping ECs among young adult dual users who are quitting CCs.

The investigators will recruit and consent 390 participants with the aim of retaining 312 (80%) by the end of treatment. Participants in each condition will complete a survey at baseline, weekly surveys throughout the 3-month treatment period, brief daily surveys for one week before and one week after the assigned quit date, an end of treatment survey, and a survey at a follow-up 6 months after treatment began. In addition, participants will provide breath CO samples at baseline, all weekly surveys, the end of treatment, and the 6-month follow-up using the CoVita iCO personal smokerlyzer (https://www.covita.net/ico-overview/).

All assessments will be remote and accessible by smartphone, tablet, or computer. After confirming eligibility and consenting to participate, participants will be randomly assigned to one of the four study groups and study personnel will mail a welcome package including study information, a CoVita iCO personal smokerlyzer device, and NRT (for groups A and B only). Upon receipt of the welcome package, participants will complete a brief baseline survey on the internet and provide a baseline breath CO sample using the CoVita iCO device and Vincere Health mobile application which is compatible with Mac iOS and Android operating systems for smartphones and tablets. The investigators will not ask participants to return their personal CoVita iCO Smokerlyzer. All participants will be free to keep their personal CoVita iCO Smokerlyzer after the conclusion of their participation.

All participants will complete brief daily surveys for two weeks: one week pre- and one week post-quit date. Participants will receive a daily text and/or email containing a link for the daily survey and will be able to complete the survey via internet on a smartphone, tablet or computer. Participants will report CC smoking, EC use, NRT use (groups A and B only), text message utilization, nicotine dependence, quit attempts, and adverse events on daily surveys (Table 2). At the conclusion of the 12-week treatment period, participants will complete an end of treatment survey to report CC smoking or EC use and withdrawal symptoms. Those still smoking will also report motivation to quit, nicotine dependence, and self-efficacy to quit. In addition, participants will provide another breath CO sample using their CoVita iCO device. The primary outcome for this RCT is CO confirmed 7-day point-prevalence abstinence from CCs at the end of treatment (i.e., at the 3-month follow-up). Per the Society for Research on Nicotine and Tobacco (SRNT) report on biochemical verification, the investigators will use CO of < 6 parts per million (ppm) as the cutoff for confirming CC abstinence. The investigators will not contact participants for the 12 weeks following the treatment period. All participants will then complete a 6-month follow-up survey (i.e., 24 weeks after the baseline assessment) to report any CC smoking or EC use and withdrawal symptoms. Those who relapsed or continued to smoke CCs will also report motivation to quit, nicotine dependence, and self-efficacy to quit. In addition, all participants will provide a final breath CO sample using their CoVita iCO device.

Treatment. The consent form explains that a primary aim of this RCT is to test whether quitting versus continuing ECs is more effective when quitting CCs, and currently there is mixed evidence supporting both strategies. After randomization, all participants will receive information about the study including instructions to set a quit date and which product(s) to quit. Written instructions for the intervention will be provided and participants will also be asked to view a supplementary video presentation. The investigators will provide participants in groups A and C with instructions to quit CCs but continue using ECs with the rationale that ongoing use of ECs could help them abstain from CCs. Specifically, the investigators will instruct participants in groups A and C to use ECs in place of CCs to help cope with cravings or urges to smoke CCs. In contrast, participants randomized to conditions B and D will receive instructions to quit CCs and quit ECs with the rationale that quitting ECs could help them abstain from CCs. The investigators will instruct participants in groups B and D to abstain from vaping because ECs could trigger relapse to CCs. Participants in groups A and B will also receive instructions for how to use NRT.

Participants randomized to conditions A and B will be mailed 3 one-month supplies of dual 14 mg NRT patches and 4 mg mini-lozenge because this appears to be the most effective non-prescription medication combination for smoking cessation However, participants will have the option to stop receiving NRT from the study. Participants will be instructed to start using both forms of NRT 2 weeks prior to their quit date because pre-quit NRT appears to increase the effectiveness of NRT. Further, the recommended use for the NRT has recently been changed to incorporate use while smoking because "the FDA has determined that there are no significant concerns with using NRT products at the same time as another nicotine-containing product like a cigarette (https://www.nicodermcq.com/faq.html)." The investigators will instruct participants to use one patch per day and use mini-lozenges when they have cravings to smoke CCs (condition A) or cravings to smoke CCs or use ECs (condition B), without surpassing 24 mini-lozenges in one 24-hour period. Anyone for whom NRT is contraindicated will be excluded from the proposed RCT. In addition, though risk of serious adverse events from NRT is low, the investigators will assess adverse events related to study procedures on nightly surveys.

All participants will receive daily text message support throughout the 12-week treatment period. The investigators will modify a text message library from SmokefreeTXT, a free interactive text message cessation service provided by Smokefree.gov that has been used with young adult smokers, uses empirically validated Behavior Change Techniques, and has been employed to support engagement in prior smoking cessation research. Data from the investigators' ongoing research indicate young adult smokers generally find daily text messages to be helpful and acceptable. The investigators will modify text messages according to participants' assigned group. For example, text messages for participants in groups A and B will encourage regular use of NRT throughout the study period. Text messages for groups B and D will support CC and EC cessation while messages for groups A and C will support CC cessation and EC continuation. The text message service will be interactive for all participants. In addition to receiving daily texts, participants will have the opportunity to send text messages to the investigators' service which will prompt automatic responses. The investigators will work with ICF incorporated, the provider for National Cancer Institute's SmokefreeTXT platform, to deliver all daily text messages and to deliver links to daily surveys.

ELIGIBILITY:
Inclusion criteria:

* Young adult
* Smokes tobacco cigarettes
* Uses electronic cigarettes
* Interested in quitting tobacco

Exclusion criteria:

* Pregnant or planning to become pregnant
* Breastfeeding or planning to start breastfeeding
* One or more contraindications for nicotine replacement therapy

Additional criteria will be assessed to determine eligibility.

If you are interested in participating, please visit the study website to find out if you are eligible: https://www.uvmquitsmokingstudy.org/

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2021-06-27 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Started | 96 | 102 | 102 | 96
Completed | 73 | 86 | 77 | 75
Not Completed | 23 | 16 | 25 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support. | Total
Number analyzed (Participants) | 96 | 102 | 102 | 96 | 396
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.8 (2.5) | 25.6 (2.8) | 26.4 (2.2) | 26.2 (2.5) | 26.0 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 50 | 52 | 209
  Male | 41 | 50 | 52 | 44 | 187
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 1 | 5
  Asian | 1 | 2 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 12 | 16 | 16 | 44
  Black or African American | 12 | 1 | 1 | 0 | 14
  White | 71 | 78 | 74 | 68 | 291
  More than one race | 10 | 7 | 8 | 9 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 16 | 11 | 55
  Not Hispanic or Latino | 82 | 88 | 86 | 85 | 341
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Confirmed 7-day Point-prevalence Cigarette Abstinence
Description: The investigators will report breath carbon monoxide (CO; <6 ppm) confirmed 7-day point-prevalence abstinence from combustible cigarettes at the end of treatment.
Time Frame: End of treatment (ie., the 3 month follow up)
Population: Breath carbon monoxide (CO) data were unavailable for the majority of participants due to a software malfunction with the app used to remotely transmit data from the CoVita iCO Smokerlyzer devices.
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 51 | 52 | 57 | 61
Participants | 16 | 26 | 16 | 16

2. Primary Outcome: Self-reported 7-day Point-prevalence Cigarette Abstinence
Description: The investigators will report self-reported 7-day point-prevalence abstinence from combustible cigarettes at the end of treatment.
Time Frame: End of treatment (ie., the 3 month follow up)
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 96 | 102 | 102 | 96
Participants | 44 | 56 | 40 | 39

3. Primary Outcome: Adverse Events During Treatment
Description: Total number of participants who reported any adverse event during the 3-month treatment period.
Time Frame: The 3 month treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 96 | 102 | 102 | 96
Participants | 7 | 11 | 8 | 12

4. Secondary Outcome: Biochemically Confirmed Prolonged 30-day Abstinence
Description: The investigators will report CO confirmed 30-day prolonged abstinence from combustible cigarettes at the 3 month follow up.
Time Frame: The 3-month follow up (ie., end of treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 51 | 52 | 57 | 61
Participants | 10 | 21 | 13 | 12

5. Secondary Outcome: Self-reported Prolonged 30-day Abstinence
Description: The investigators will report self-reported 30-day prolonged abstinence from combustible cigarettes at the 3- and 6-month follow ups.
Time Frame: The 3-month follow up (ie., end of treatment) and 6-month follow up (3 months after the end of treatment).
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 96 | 102 | 102 | 96
Participants
  3-month follow-up | 27 | 48 | 31 | 28
  6-month follow-up | 44 | 43 | 38 | 41

6. Secondary Outcome: Any Attempts to Quit Combustible Cigarettes
Description: The investigators will report the percent of participants who made a quit attempt lasting any length of time (including very short quit attempts) during treatment.
Time Frame: The 3-month treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 96 | 102 | 102 | 96
Participants | 89 | 100 | 92 | 88

7. Secondary Outcome: Cigarettes Per Day
Description: The investigators will report cigarettes per day during the 3 month treatment period among participants who continue to smoke cigarettes.
Time Frame: The 3-month treatment period.
Population: This analysis is limited to the subset of participants who reported continued smoking at the 3-month follow-up.
Measure: Mean (Standard Deviation); unit: Cigarettes per day during the prior week
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 29 | 30 | 37 | 33
Cigarettes per day during the prior week | 4.67 (6.05) | 4.67 (4.75) | 4.37 (5.32) | 4.84 (5.37)

8. Secondary Outcome: Cigarette Dependence
Description: The investigators will report cigarette dependence using the Patient Reported Outcomes Measurement Information System (PROMIS) measure of cigarette dependence (total score of 0=least to 4=most dependent) during the 3 month treatment period among participants who continue to smoke cigarettes.
Time Frame: The 3-month treatment period.
Population: This analysis is limited to the subset of participants who reported continued smoking at the 3-month follow-up.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
Number analyzed (Participants) | 29 | 30 | 37 | 33
Scores on a scale | 1.78 (1.30) | 1.71 (1.14) | 1.58 (1.10) | 1.70 (1.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 3-month treatment period.
Description: All participants were asked if they experienced one or more adverse events on each weekly survey during the 3-month treatment period.
Arm/Group | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. | Quit Cigarettes and Quit E-cigarettes With Text Support.
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/102 | 0/102 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/102 | 0/102 | 0/96
Other Adverse Events (participants affected / at risk) | 7/96 | 11/102 | 8/102 | 12/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quit Cigarettes, But Continue Using E-cigarettes, With Nicotine Replacement Therapy and Text Support (N=96) | Quit Cigarettes and Quit E-cigarettes With Nicotine Replacement Therapy and Text Support. (N=102) | Quit Cigarettes, But Continue Using E-cigarettes, With Text Support. (N=102) | Quit Cigarettes and Quit E-cigarettes With Text Support. (N=96)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pregnancy, pueperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 2 (3) | 9 (9) | 4 (4) | 7 (7)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04946825/Prot_SAP_000.pdf